CLINICAL TRIAL: NCT02120339
Title: Beta Blockers in Pulmonary Arterial Hypertension (PAH) A Pilot Study of Efficacy and Safety
Brief Title: Carvedilol PAH A Pilot Study of Efficacy and Safety
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PAH
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Pulmonary Hypertension; Cardiac MRI <40
Keywords: Hypertension; PAH
MeSH Terms: conditions — Hypertension, Pulmonary; Hypertension | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carvedilol (Experimental): Carvedilol 0-3.125 mg daily Escalating to 6.25 twice a day
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol

SUMMARY:
Estimate the effect of chronic beta-adrenergic receptor blockade with carvedilol on RV function in patients with PAH.

Assess the safety and tolerability of chronic carvedilol therapy in patients with PAH

DETAILED DESCRIPTION:
This is a prospective, open label, uncontrolled, pilot study examining the safety and efficacy of beta-blocker therapy with carvedilol on RV function in stable PAH Patients with World Health Organization (WHO) functional class II or III symptoms and RV ejection fraction (EF) < 40%. Twenty-five evaluable patients will be enrolled at the University of Minnesota.

Specific Aims:

1.1 Primary Efficacy Endpoint: Adult males and females on a stable dose of an approved PAH medication will undergo cardiac magnetic resonance imaging (MRI), right heart catheterization (RHC), echocardiogram, 6-minute walk test (6-MWT), measurement of plasma NT-ProBNP and serum catecholamine, and quality of life assessment. Patients will receive carvedilol (3.25 mg/kg bid escalating to 25 mg/kg bid over 3 months). Testing is repeated at the end of the study (month 6). RVEF measured by cardiac MRI is the primary efficacy endpoint. We define a 5% increase in RVEF as a meaningful change.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be eligible to participate in the study if all of the following conditions exist:
2. Age > 18 years
3. WHO category 1 pulmonary arterial hypertension (Dana Point 2008)
4. WHO functional class II-III
5. RVEF by cardiac MRI < 40%
6. Mean pulmonary artery pressure > 40 mm Hg
7. Stable on PAH-specific therapy as defined by no change in PAH-specific treatment and functional class in the past 3 months. Patient can be on either mono or combination PAH-specific therapy

Exclusion Criteria:

* 1. Subjects will be excluded from participation in the study if any of the following conditions exist: 2. Significant persistent bradycardia (resting heart rate < 60 bpm) without a permanent pacemaker 3. Second or third degree AV block without a permanent pacemaker 4. Significant sinus tachycardia (resting heart rate > 100 bpm) 5. Use of anti-arrhythmic drugs 6. Hypotension defined as systolic blood pressure < 100 mmHg at the time of enrollment 7. Significant illness in the past 30 days requiring hospitalization 8. Acute decompensated right heart failure within past 30 days 9. Known allergy or intolerance to carvedilol or other β blockers 10. Cardiac index < 2 l/min/m2 or right atrial pressure > 15 mm Hg 11. Asthma

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean change in RVEF | Baseline and 6 months
  1. The primary efficacy outcome is the mean change in RVEF as measured by cardiac MRI before and after 6 months of carvedilol treatment. An improvement of 5% will be considered to be clinically significant. Assessment of the RV is challenging due to its complex geometry. Cardiac MRI offers the ability to acquire 3-dimensional datasets that do not require geometric modeling. In addition to being highly reproducible40, RVEF measured by cardiac MRI can be used to identify PAH patients that are likely to have clinical worsening41. The prognostic ability of cardiac MRI-measurements of RVEF is similar to that as mean pulmonary artery pressure and exercise capacity

SECONDARY OUTCOMES:
Absence of Adverse Events | 6 months
  The primary safety outcome is the absence of adverse events associated with carvedilol including hypotension (<90 mm Hg), bradycardia (<50 bpm or advanced atrioventricular nodal block), bronchospam, or acute decompensated right heart failure requiring hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Thenappan Thenappan, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Thenappan T, Weir EK, Prins KW, Pritzker MR, Archer SL. Carvedilol for Treatment of Right Ventricular Dysfunction in Pulmonary Arterial Hypertension. J Am Heart Assoc. 2021 Jul 20;10(14):e021518. doi: 10.1161/JAHA.121.021518. Epub 2021 Jul 14. No abstract available. PMID 34259020